CLINICAL TRIAL: NCT02749916
Title: Contrast Enhanced Susceptibility Weighted Imaging (SWI) for Characterization of Carotid Plaque
Brief Title: Contrast Enhanced SWI for Carotid Plaque Imaging
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hyun Seok Choi, M.D. (Other)
Responsible Party: Sponsor-Investigator, Hyun Seok Choi, M.D., Associate professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: KC15EIMI0104
Record Dates: First submitted 2016-04-19; First posted 2016-04-25 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Carotid Plaque Imaging
Keywords: SWI; MP-RAGE; DANTE T1-SPACE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute or recent (within 3months) stroke
  Interventions: Other: Methods of carotid wall imaging

INTERVENTIONS:
Other: Methods of carotid wall imaging

SUMMARY:
This study aims to compare image-based characteristics of carotid walls between symptomatic side and the opposite side. The design of this study is phase IV, prospective observational study.

DETAILED DESCRIPTION:
Atherosclerosis of craniocervical arteries are one of most important causes of stroke. Carotid artery is the most frequent site of atherosclerosis. Recent research in carotid artery covers not only morphology of lumen but also direct visualization of carotid plaque or vessel wall. Vulnerable carotid plaques share pathologic features of intra-plaque inflammation and hemorrhage. There have been reports about post-contrast SWI in the field of vascular imaging. We hypothesized SWI is so sensitive to gadolinium based contrast agent and hemorrhage that contrast-enhanced SWI can visualize vulnerable carotid plaque. The purpose of this study is to investigate gadolinium-enhanced SWI in detection of vulnerable carotid plaque and compare it with MP-RAGE and DANTE T1-SPACE. This can be used to guide proper treatment for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or recent (within 3months) stroke or TIA
* 50-99% stenosis of internal carotid artery by NASCET criteria
* Written informed consent, prior to registration

Exclusion Criteria:

* Hemorrhagic stroke
* Previous history of carotid endarterectomy (CEA), angioplasty, or stenting
* Contraindication for MR imaging
* Hypersensitivity to gadolinium based contrast media
* Pregnant or lactating women
* Patients under age of 19-year-old
* Renal condition : eGFR < 60
* Patients unable and/or unwilling to comply with treatment or study instructions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or recent (within 3months) stroke or TIA (transient ischaemic attack)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of findings of vulnerable carotid plaque | within 3 days after enrollment

SECONDARY OUTCOMES:
Accuracy in delinating geometry of carotid inner lumen and outer wall | within 3 days after enrollment
  Diameter of inner lumen and outer wall; Area of inner lumen and outer wall

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No